CLINICAL TRIAL: NCT01243216
Title: The Utility of Pre-procedure Ultrasound for Neuraxial Analgesia/Anesthesia in Obstetric Patients
Brief Title: Does Ultrasound of the Spine Improve Labor Epidurals/Spinal Anesthesia in Obstetric Patients?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of personnel/research time
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1167437
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Pregnancy; Labor Pain
Keywords: Pregnancy; Labor; Epidural Analgesia; Epidural Anesthesia; Spinal Anesthesia; Ultrasound; Neuraxial Analgesia; Neuraxial Anesthesia; Cesarean delivery
MeSH Terms: conditions — Labor Pain | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound Group (Experimental): Patients in the Ultrasound Group will have a pre-procedure ultrasound of the spine prior to needle placement
  Interventions: Device: Ultrasound
- No Ultrasound Group (No Intervention): Patients in the No Ultrasound Group will not have a pre-procedure ultrasound of the spine performed prior to needle placement.

INTERVENTIONS:
Device: Ultrasound — Ultrasound examination of the lumbar spine. The level of the lumbar interspace will be determined by the oblique/sagittal method. The transverse method will be used to determine the best lumbar interspace and the distance from the skin to the target (epidural space or intrathecal space)
  Arms: Ultrasound Group

SUMMARY:
The investigators are interested in determining the utility of ultrasound of the spine for labor epidurals or spinal anesthesia for women in labor or having a cesarean delivery. The investigators hypothesized that in women with poor spinal landmarks that the use of ultrasound of the spine will improve the process of placing labor epidurals or spinal anesthetics

DETAILED DESCRIPTION:
Ultrasound has been in use for peripheral regional anesthesia for several years and is becoming more common. It is currently routinely used here at the University of Missouri. Ultrasound for neuraxial anesthesia, however, is less common and is only being done in a few centers.. There have been several case reports of its use in obstetric anesthesia for patients with prior spinal surgery or spinal deformity. There have been even few prospective randomized studies. While its use may have significant advantages, it is not yet clear what those advantages are and in whom it may be most beneficial. The investigators seek to answer the following questions regarding the use of preprocedure ultrasound for neuraxial analgesia/anesthesia in obstetric patients:

* Are there benefits to the use of pre procedure ultrasound for neuraxial analgesia/anesthesia?
* If so, what are the benefits?
* If measurable, to what extent does the patient benefit?
* Do all patients benefit or only a specific subgroup?
* Is there a "cost" to the use of pre procedure ultrasound, i.e. extra time needed to perform the ultrasound exam vs a "savings" with the use of pre procedure ultrasound, i.e., less time to perform the epidural analgesic or spinal anesthetic as a direct result of the use of ultrasound?
* In particular the investigators hypothesize that in patients whose spinal landmarks are not palpable or are barely palpable, ultrasound will be found to be beneficial as determined by metrics described below (see item #6). In patients whose landmarks are prominent or easily palpable pre procedure ultrasound will not be of significant benefit.

ELIGIBILITY:
Inclusion Criteria:

* Women in labor
* Women scheduled for cesarean delivery

Exclusion Criteria:

* Under age 18
* Emergency cesarean deliveries
* Unable to cooperate with ultrasound examination or regional anesthesia
* Advanced labor
* Contraindications to regional anesthesia
* Unable to understand the consent process

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of attempts needed for proper needle placement | 30 min or less
  An attempt is defined as a separate needle puncture. A needle pass is defined as the passage of a needle through a single puncture site

SECONDARY OUTCOMES:
Time | 30 min
  The time for performance of an ultrasound exam as well as the time for needle placement for labor epidurals or spinal anesthesia
Patient Satisfaction | 30 min
  Patients will be given a questionaire grading their satisfaction on a 1 to 5 scale 1-very unsatisfied, 5-very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Steven T Fogel, M.D., Principal Investigator — University of Missouri-Columbia School of Medicine
Locations (1):
- Women's and Children's Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvalho JC. Ultrasound-facilitated epidurals and spinals in obstetrics. Anesthesiol Clin. 2008 Mar;26(1):145-58, vii-viii. doi: 10.1016/j.anclin.2007.11.007. PMID 18319185
- [Background] Arzola C, Davies S, Rofaeel A, Carvalho JC. Ultrasound using the transverse approach to the lumbar spine provides reliable landmarks for labor epidurals. Anesth Analg. 2007 May;104(5):1188-92, tables of contents. doi: 10.1213/01.ane.0000250912.66057.41. PMID 17456672
- [Background] Chin KJ, Perlas A, Singh M, Arzola C, Prasad A, Chan V, Brull R. An ultrasound-assisted approach facilitates spinal anesthesia for total joint arthroplasty. Can J Anaesth. 2009 Sep;56(9):643-50. doi: 10.1007/s12630-009-9132-8. Epub 2009 Jun 23. PMID 19548051
- [Background] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Background] Grau T, Leipold RW, Conradi R, Martin E. Ultrasound control for presumed difficult epidural puncture. Acta Anaesthesiol Scand. 2001 Jul;45(6):766-71. doi: 10.1034/j.1399-6576.2001.045006766.x. PMID 11421838